CLINICAL TRIAL: NCT01674933
Title: Comparison Of The Caries-Protective Effect Of Fluoride Varnish (Duraphat®) With Treatment As Usual In Nursery School Attendees Receiving Preventive Oral Health Support Through The Childsmile Oral Health Improvement Programme: An RCT
Brief Title: Fluoride Varnish For Childsmile Nursery School Attenders
Acronym: PT@3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: NHS Research Scotland (Other)
Responsible Party: Principal Investigator, Lorna Macpherson, Professor, Glasgow Dental School, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GC12CO201
Record Dates: First submitted 2012-08-24; First posted 2012-08-29 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Dental Caries
Keywords: dental; prevention; caries; oral; children
MeSH Terms: conditions — Dental Caries | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment as usual (Active Comparator): any treatment from the family dentist, plus the preventive intervention programme offered to nursery school children, including daily supervised toothbrushing
  Interventions: Behavioral: treatment as usual
- Duraphat® Fluoride Varnish (Experimental): treatment as usual (ie any treatment from the family dentist, plus the preventive intervention programme offered to nursery school children, including daily supervised toothbrushing) plus up to 4 six-monthly applications of Duraphat Fluoride Varnish in the nursery school setting.
  Interventions: Drug: Duraphat® Fluoride Varnish

INTERVENTIONS:
Drug: Duraphat® Fluoride Varnish — 0.25 ml per application will be painted on tooth surfaces by a Childsmile trained Extended Duties Dental Nurse, currently registered with the UK General Dental Council
  Other Names: Duraphat® Fluoride Varnish (Colgate-Palmolive).
  Arms: Duraphat® Fluoride Varnish
Behavioral: treatment as usual — includes supervised toothbrushing, distribution of toothbrushes and toothpaste and oral health advice given at nursery school.
  Arms: treatment as usual

SUMMARY:
The study will compare the effectiveness of Duraphat® fluoride varnish in preventing any further dental decay among 3-4 year old children in nursery schools.

It is important to ascertain the additional preventive value that fluoride varnish may provide when applied in conjunction with other preventive measures which form part of a national dental health improvement programme targeting children at risk from dental decay. 1600 children will be recruited into the study for 2 years.

DETAILED DESCRIPTION:
The objective of this study is to compare the effectiveness of Duraphat® fluoride varnish plus treatment as usual (TAU) with TAU only in preventing any further dental decay.

Thus the study is a clinical trial of treatment as usual (TAU) versus TAU plus fluoride varnish in the nursery school setting. TAU is the core Childsmile Nursery intervention (supervised daily toothbrushing with fluoride toothpaste, free dental packs of fluoride toothpaste, toothbrushes and advice).

Children will be screened by asking parents whether or not the child has previously been hospitalised with asthma or diagnosed with any allergies. Provided that a child has no contraindications to fluoride varnish then the child can proceed to study inclusion. On the day of the planned application, the dental nurse will carry out a risk assessment to reduce the possibility of children with oral/facial infections being included. After excluding non-eligible children, a baseline dental examination will take place, followed by randomisation into treatment as usual or treatment as usual plus fluoride varnish. This second group will receive up to four fluoride varnish applications at 6 month intervals. After two years, all study children will be offered a final dental examination.

ELIGIBILITY:
Inclusion Criteria:

* Children attending nurseries which cover significant numbers of children whose home postcode is within the most deprived quintile of postcodes as measured by the Scottish Index of Multiple Deprivation (SIMD) (Scottish Government 2011).
* Children in the first year of nursery school (known as the 'ante pre school year'). On average the children will be three years old.
* Every eligible child in participating nurseries will be invited to join the study, irrespective of the SIMD ranking of their own postcode.
* Children with or without pre-existing cavities, as the cavity can be treated through the usual primary care dental service (i.e. as part of 'treatment as usual').

Exclusion Criteria:

* Children with contraindications for the Duraphat® varnish i.e. hypersensitivity to colophony and/or any other constituents, ulcerative gingivitis, stomatitis, bronchial asthma, history of allergic episodes requiring hospital admission (e.g. asthma).
* Receipt of fluoride supplements due to a small risk of fluorosis.
* Abnormalities of the skin around the mouth, lips (e.g. cold sores) and soft tissue lesions.

Ages: 36 Months to 50 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1610 (Estimated)
Dates: Start 2012-10; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
d3mft ( a standard measure of dental health (number of teeth where decay which has penetrated the tooth enamel, plus the number of missing or filled teeth) | 24 months
  d3mft is a standard measure of dental health (number of teeth where decay which has penetrated the tooth enamel, plus the number of missing or filled teeth).

SECONDARY OUTCOMES:
d3mfs | 24 months
  a standard measure of dental health, comprising the number of tooth surfaces where decay which has penetrated the tooth enamel, plus the number of missing or filled teeth

OTHER OUTCOMES:
child oral quality of life | 24 months
  quality of life using a disease specific questionnaire designed by the University College London. Cost effectiveness will be expressed as cost per quality adjusted life years (QALYs). The economic analysis will estimate the mean costs and QALYs, with standard deviations or standard errors or as mean differences with 95% confidence intervals, over two years in the first instance.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna MD Macpherson, Principal Investigator — University of Glasgow
Locations (4):
- United Kingdom (4):
  - NHS Lothian, Edinburgh, Scotland
  - NHS Greater Glasgow and Clyde, Glasgow, Scotland
  - NHS Fife, Kirkcaldy, Scotland
  - NHS Tayside, Perth, Scotland

REFERENCES:
- [Derived] Wright W, Turner S, Anopa Y, McIntosh E, Wu O, Conway DI, Macpherson LM, McMahon AD. Comparison of the caries-protective effect of fluoride varnish with treatment as usual in nursery school attendees receiving preventive oral health support through the Childsmile oral health improvement programme - the Protecting Teeth@3 Study: a randomised controlled trial. BMC Oral Health. 2015 Dec 18;15:160. doi: 10.1186/s12903-015-0146-z. PMID 26681191